CLINICAL TRIAL: NCT05252988
Title: A Randomized Phase II Study to Evaluate the Incidence of Discontinuations Due to Diarrhoea at 3 Cycles in Patients With Early-stage HER2-positive (HER2+), Hormone Receptor-positive (HR+) Breast Cancer Treated With Neratinib Plus Loperamide Prophylaxis Versus Neratinib With Initial Dose Escalation Plus PRN Loperamide Prophylaxis Versus Neratinib Plus Loperamide Plus Colesevelam Prophylaxis "DIANER Study"
Brief Title: Three Antidiarrheal Strategies in HER2+/HR+ Early Breast Cancer Patients Treated With Extended Adjuvant Neratinib
Acronym: DIANER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Puma Biotechnology, Inc. (Industry); Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GEICAM/2018-06; 2019-001559-38 (EudraCT Number)
Record Dates: First submitted 2022-02-02; First posted 2022-02-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Early-stage Breast Cancer; HER2 Positive Breast Cancer; Hormone Receptor Positive
Keywords: Early-stage Breast Cancer; HER2 positive; Hormone Receptor positive; Neratinib; Loperamide prophylaxis; Colesevelam prophylaxis; Incidence of Discontinuations due to Diarrhoea
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Loperamide; Colesevelam Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): 1. Neratinib 240 mg (six 40mg tablets) orally once daily for 13 cycles (C) (1 C = 28 days), unless patient discontinues earlier.
  2. Mandatory loperamide 4 mg (2 tablets/capsules) orally, 3 times a day (total 12 mg a day) starting Day (D) 1 of neratinib and for the first 14 days. Then, 4 mg (2 tablets/capsules) orally, 2 times a day (total 8 mg a day) until the end of C2 (D56); thereafter, loperamide will be administered PRN (without exceeding 16 mg per day).
  Interventions: Drug: Neratinib; Drug: Loperamide
- Arm B (Experimental): 1. Neratinib 120 mg for Week 1 (C1D1 - C1D7), followed by 160 mg neratinib for Week 2 (C1D8 - C1D14), followed by 240 mg neratinib for Week 3 and thereafter for 13 cycles inclusive, until cycle 13 day 28 (unless patient discontinues earlier).
  2. Loperamide to be administered PRN only (without exceeding 16 mg per day).
  Interventions: Drug: Neratinib; Drug: Loperamide
- Arm C (Experimental): 1. Neratinib 240 mg (six 40-mg tablets) orally once daily for 13 C, unless patient discontinues earlier.
  2. Mandatory loperamide 4 mg (2 tablets/capsules) orally, 3 times a day (total 12 mg a day) for the first 14 days. After the first 14 days, 4 mg (2 tablets/capsules) orally, 2 times a day (total 8 mg a day) to complete a total of 28 days.
  3. Mandatory colesevelam 1,875 mg (three 625-mg capsules orally), 2 times a day for the first month (28 days). After day 28, any prophylaxis or treatment for diarrhoea could be administered PRN, if loperamide not to exceed 16 mg per day.
  Interventions: Drug: Neratinib; Drug: Loperamide; Drug: Colesevelam

INTERVENTIONS:
Drug: Neratinib — Neratinib orally once daily for 13 cycles, unless patient discontinues earlier.
  Other Names: Nerlynx
Drug: Loperamide — Loperamide orally.
  Other Names: Sindiar
Drug: Colesevelam — Colesevelam capsules orally, 2 times a day for the first month (28 days).
  Other Names: Cholestagel
  Arms: Arm C

SUMMARY:
A Randomized Phase II Study to Evaluate the Incidence of Discontinuations due to Diarrhoea at 3 Cycles in patients with Early-stage HER2-positive (HER2+), Hormone Receptor-positive (HR+) Breast Cancer treated with Neratinib plus Loperamide prophylaxis versus Neratinib with Initial Dose Escalation plus PRN Loperamide prophylaxis versus Neratinib plus Loperamide plus Colesevelam prophylaxis.

DETAILED DESCRIPTION:
This is an international, multicenter, prospective, controlled, randomized, adaptative, phase II study to evaluate the incidence of discontinuations due to diarrhoea within the first 3 cycles in patients with early-stage HER2+ and HR+ breast cancer treated with neratinib plus loperamide prophylaxis for the first 2 cycles versus neratinib with initial 2-week dose escalation plus PRN loperamide versus neratinib and loperamide plus colesevelam prophylaxis for 28 days.

After the preplanned therapy, prophylaxis or treatment for diarrhoea will be given as clinically indicated following the standard of care by the treating physician.

Approximately 315 patients will be enrolled in the study.

All enrolled patients will receive neratinib orally once daily for 13 cycles, continuously. Eligible patients will be randomly assigned in a 1:1:1 ratio to one of the diarrhoea prophylaxis arms, using an interactive response technology (IRT) module within the electronic data capture (EDC) system. Patients will be stratified according to menopausal status (premenopausal versus postmenopausal) and prior anti-HER2 therapy (trastuzumab only versus trastuzumab plus pertuzumab).

Baseline assessments will be performed prior to C1D1 dosing. During the first 3 cycles of treatment, safety data will be collected during the cycle visits. After the first 3 cycles, all patients will enter in a follow-up period to complete approximately 1 year of neratinib treatment. During this follow-up period, safety data will be collected every 3 months. An End-of-Treatment (EOT) Visit is planned on cycle 13 day 28 for all treatment arms (unless patient discontinues earlier), followed by a Safety Follow-up Visit (30 +/-5 days after the last dose of neratinib). This will be the core phase of the study.

After this safety follow-up visit, long term outcome data will be collected for 5 years to address the exploratory objectives. This will be the extended phase of the study. Archived primary tumor tissue (at baseline) and whole blood samples (at baseline, during the treatment and follow-up period, and at disease relapse) will be collected for the exploratory analyses.

Patients are anticipated to participate in the core phase of the study for approximately 1 year to address primary and secondary objectives (28 days for screening, approximately 12 months to complete neratinib treatment, and 30 days for a safety follow-up visit after the last dose of neratinib). Later on patients will continue in the extended phase of the study and will be followed-up for at least 5 years to collect long term outcome data to conduct the exploratory analyses. The approximate duration of the full study is 8 years.

The objectives of the study are indicated below:

Primary objectives:

To evaluate the incidence of neratinib discontinuations due to diarrhoea within the first 3 cycles (1 cycle = 28 days) in patients with early-stage HER2 overexpressed/amplified (HER2+), hormone receptor-positive (HR+) breast cancer who have completed adjuvant trastuzumab-based therapy.

Primary End-point:

Incidence of neratinib discontinuations due to diarrhoea at the end of 3 cycles of neratinib treatment.

Secondary Objectives:

* Incidence and time of neratinib discontinuations due to any treatment-emergent adverse event (TEAE).
* Diarrhoea due to neratinib: incidence, duration, severity, and treatment interventions.
* Incidence of neratinib discontinuation due to any reason.
* Incidence of hospitalisations (overall and for diarrhoea).
* Incidence of TEAEs and serious adverse events (SAEs) and adverse events of special interest (AESIs, ie, hepatic, cardiac, pulmonary, reproductive and developmental).
* Neratinib exposure assessment.
* Determine the effect of study treatment on quality of life, as measured by patient reported outcomes, in all treatment arms.

Secondary End-points:

* Incidence and time to neratinib discontinuations due to any TEAE.
* Incidence, cumulative duration and time to first episode of any diarrhoea and grade 3 or higher diarrhoea.
* Incidence and time to neratinib discontinuation due to any reason.
* Incidence of hospitalisations due to any reason and diarrhoea.
* Incidence of TEAEs and SAEs that included AESIs (i.e. hepatic, cardiac, pulmonary, reproductive and developmental).
* Incidence of Neratinib dose modifications (reductions and dose holds), and dose intensity.
* Systemic therapy-induced diarrhea Assessment Tool (STIDAT), Functional Assessment of Cancer Therapy Questionnaire for Breast Cancer (FACT B) and EuroQol 5 Dimensions 5 Levels (EQ5D-5L) questionnaires.

Exploratory Objectives:

Evaluate minimal residual disease (MRD) and molecular alterations associated with patient outcome, and/or the development of diarrhoea with neratinib.

Exploratory End-points:

Correlation of biomarkers data with patient outcome and safety data.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be enrolled in the study only if they meet all of the following criteria:

1. Male or female patient ≥18 years of age at signing of informed consent.
2. Histologically confirmed Stage I B through Stage III C primary adenocarcinoma of the breast.
3. Documented HER2-positive disease based on local laboratory determination according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) 2018 criteria.
4. Documented HR+ disease, defined as oestrogen receptor (ER) and/or progesterone receptor (PR) ≥1% based on local laboratory determination.
5. Patients must have completed prior neoadjuvant/adjuvant trastuzumab-based therapy (eg, trastuzumab-based treatments including trastuzumab-emtansine [T-DM1]) or experienced side effects that resulted in early discontinuation of trastuzumab-based therapy that have since resolved (pertuzumab therapy is accepted but not mandatory).
6. The last dose of trastuzumab-based therapy must have been given to the patient >2 weeks and ≤1 year (365 days) before first dose of neratinib.
7. Left ventricular ejection fraction (LVEF) ≥50% measured by multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO).
8. Eastern Cooperative Oncology Group (ECOG) status of 0 or 1.
9. Negative β-human chorionic gonadotropin (hCG) pregnancy test for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after menopause. [Women are considered postmenopausal if they are ≥ 12 months without menses, in the absence of endocrine or anti-endocrine therapies].
10. Women of childbearing potential must agree and commit to the use of a highly effective non-hormonal method of contraception, ie, intrauterine device, bilateral tubal ligation, vasectomized partner, or abstinence (only when it is the preferred lifestyle of the patient), from the time of informed consent until 30 days after the last dose of the medicinal products. Male patient with female partner of childbearing potential must agree and commit to use condom, and the female partner must agree and commit to use a highly effective method of contraception (ie, any of the above methods, or for females, hormonal contraception associated with inhibition of ovulation) while on treatment and for 3 months after last dose of medicinal products.
11. Recovery (ie, to Grade 1 or baseline) from all clinically significant AEs related to prior therapies (excluding alopecia, neuropathy, and nail changes).
12. Provide written, informed consent to participate in the study and follow the study procedures.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Clinical or radiologic evidence of local or regional recurrence of disease or metastatic disease prior to or at the time of study entry.
2. Currently receiving chemotherapy, radiation therapy, immunotherapy, or biological therapy for breast cancer (adjuvant endocrine therapy is allowed).
3. Major surgery within <30 days of starting treatment or received chemotherapy, investigational agents, or other cancer therapy <14 days prior to the initiation of investigational products.
4. Active uncontrolled cardiac disease, including cardiomyopathy, congestive heart failure (New York Heart Association functional classification of ≥2), unstable angina, myocardial infarction within 12 months of enrolment, or ventricular arrhythmia.
5. Corrected QT interval (QTc) interval >0.450 seconds (males) or >0.470 (females), or known history of QTc prolongation or Torsade de Pointes (TdP).
6. Screening laboratory assessments outside the following limits:

   Absolute neutrophil count (ANC) ≤1,000/μl (≤1.0 x 109/L), Platelet count ≤100,000/μl (≤100 x 109/L), Hemoglobin ≤9 g/dL, Total bilirubin >1.5 x institutional upper limit of normal (ULN) (in case of known Gilbert's syndrome, <2 x ULN is allowed), Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x institutional ULN, Creatinine clearance <30 mL/min (as calculated by Cockcroft-Gault formula a or Modification of Diet in Renal Disease (MDRD) formula).
7. Active, unresolved infections.
8. Patients with a second malignancy, other than adequately treated non-melanoma skin cancers, in situ melanoma or in situ cervical cancer. Patients with other non-mammary malignancies must have been disease-free for at least 5 years.
9. Currently pregnant or breast-feeding.
10. Significant chronic gastrointestinal disorder with diarrhoea as a major symptom (eg, Crohn's disease, malabsorption, or Grade ≥2 National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events Version 5.0 [CTCAE v.5.0] diarrhoea of any etiology at baseline); or gastroparesis, dysphagia, or swallowing disorder.
11. Clinically active infection with hepatitis B or hepatitis C virus.
12. Evidence of significant medical illness, abnormal laboratory finding, or psychiatric illness/social situations that could, in the Investigator's judgment, make the patient inappropriate for this study.
13. Known hypersensitivity to any component of the investigational products; known allergies to any of the medications or components of medications used in the trial.
14. Unable or unwilling to swallow tablets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of neratinib discontinuations due to diarrhoea at the end of 3 cycles (1 cycle= 28 days) of neratinib treatment. | Up to 3 months
  The proportion of patients who discontinue the treatment with neratinib due to diarrhoea within this time period.

SECONDARY OUTCOMES:
Incidence of neratinib discontinuations due to any TEAE (treatment-emergent adverse event). | Up to 13 months
  The proportion of patients who discontinue the treatment of neratinib at any time due to any TEAE. TEAE are undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment.
Time to neratinib discontinuations due to any TEAE (treatment-emergent adverse event). | Up to 13 months
  The time from the start of neratinib therapy to the discontinuation due to any TEAE.
Incidence of diarrhoea of any grade/grade 3 or higher. | Up to 13 months
  The proportion of patients with at least one TEAE of diarrhoea of any grade/grade 3 or higher coded and graded by the investigator according to the NCI-CTCAE version 5.0.
Cumulative duration of diarrhoea (Grade 2/3/4). | Up to 13 months
  The time from the diagnosis of each of the different diarrhoea Grades 2 or 3 or 4 coded and graded by the investigator according to the NCI-CTCAE version 5.0 to the time of change to a different grade of this adverse event.
Time to first episode of diarrhoea. | Up to 13 months
  The time from the start of neratinib therapy to the first episode of diarrhoea of any grade, whichever occurs first.
Incidence of neratinib discontinuation (for any reason). | Up to 13 months
  The proportion of patients who discontinued neratinib early (before 1 year of therapy).
Time to neratinib discontinuation/neratinib treatment duration. | Up to 13 months
  The time from the start of neratinib to the last dose of neratinib.
Incidence of hospitalisations due to any reason and diarrhoea. | Up to 13 months
  The proportion of patients who have a hospitalisation during the treatment with neratinib or 30 days after the last dose.
Incidence of TEAEs and SAEs that include AESIs (ie, hepatic, cardiac, pulmonary, reproductive and developmental). | Up to 13 months
  The proportion of patients in which those events are observed.
Cumulative dose of neratinib. | Up to 13 months
  The total dose of neratinib administered during the study.
Neratinib dose intensity. | Up to 13 months
  The cumulative dose of neratinib divided by the neratinib treatment duration.
Neratinib relative dose intensity. | Up to 13 months
  The dose intensity divided by 240 mg.
Patient reported outcomes (PRO) of health related quality of life measured by FACT B. | Up to 13 months
  PRO of health related quality of life will be assessed using the FACT-B questionnaire.
  The FACT-B is a 36-item questionnaire composed of five multi-item functional subscales: physical well-being, social/family well-being, emotional well-being, functional well-being and a subscale related with the breast cancer and its treatment. The questionnaire employs 5 points Likert scales with responses from "not at all" to "very much". The total score is obtained from the sum of the score on each subscale.
  Patients will complete a questionnaire at cycle 1 day 1 (before the first dose of neratinib and anti-diarrhoeal therapy), on day 1 of cycles 2, 3, 4, 7 and 10 and at the End of Treatment Visit.
Patient reported outcomes (PRO) of health related quality of life measured by EQ5D-5L | Up to 13 months
  To be assessed using the EQ5D-5L questionnaire, a standardized instrument for measuring generic health status. It has 2 components:
  * health state description: measured in terms of 5 dimensions; mobility (person's walking ability), self-care (ability to wash or dress by oneself), usual activities (work, study, housework, family or leisure activities), pain/discomfort (how much pain or discomfort they have), and anxiety/depression (how anxious or depressed they are). The number of levels of severity is 5; having no problems, slight problems, moderate problems, severe problems and being unable to do/extreme problems. The respondents self-rate their level of severity for each dimension.
  * Evaluation: It also includes a visual analogue scale, EQ VAS, which records patient's self-rated health on a scale from 0 (worst imaginable) to 100 (best imaginable).
  To be completed at day 1 of cycles 1, 2, 3, 4, 7 and 10 and at the End of Treatment Visit.
Patient reported outcomes (PRO) of health related quality of life measured by Systemic Therapy-Induced Diarrhea Assessment Test (STIDAT) | Up to 13 months
  PRO of health related quality of life will be assessed using the STIDAT questionnaire.
  The STIDAT is a questionnaire that was developed using the FDA iterative process for patient-reported outcomes in which patients define diarrhoea based on presence of watery stool. The STIDAT assess patient's perception of having diarrhoea, daily number of bowel movements, daily number of diarrhoea episodes, antidiarrheal medication use, the presence of urgency, abdominal pain, abdominal spasms or fecal incontinence, patient's perception of diarrhoea severity, and QoL.
  Patients will complete the instrument at cycle 1 day 1 (before the first dose of neratinib and anti-diarrhoeal therapy), on day 1 of cycles 2, 3, 4, 7, 10 and at the End of Treatment Visit.

OTHER OUTCOMES:
Minimal residual disease (MRD) | Up to 13 months
  Correlation of biomarkers data with patient outcome and safety data These analysis will be performed in the biomarker population. Given a relapse rate of around 10%, we anticipate that approximately 150-200 patients would be sufficient to explore the prognostic value of the MRD assessed on circulating tumor DNA and the correlation of the molecular and clinical relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Study Director, Study Director — Hospital General Universitario Gregorio Marañón; Study Director Study Director, Study Director — Insititut Català d'Oncologia de L'Hospitalet
Locations (55):
- Spain (55):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Costa del Sol, Málaga, Andalusia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Institut Català d'Oncología (ICO) L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Althaia Xarxa Asistencial de Manresa, Manresa, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castellón
  - Hospital Clínico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital Universitario Puerta del Mar, Cadiz, Cádiz
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Centro Oncologico de Galicia, A Coruña, Galicia
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Universitario Infanta Cristina, Parla, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario San Joan de Reus, Reus, Tarragona
  - Hospital General Universitario Dr. Balmis, Alicante, Valencia
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - OSI Barrualde-Galdakao (Hospital Galdakao-Usansolo), Usansolo, Vizcaya
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Compejo Hospitalario Universitario de Albacete, Albacete
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital Universitario Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Basurto, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario San Pedro de Alcántara, Cáceres
  - Institut Català d'Oncología (ICO) Girona, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Clínico San Cecilio, Granada
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora De Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Quirónsalud Sagrado Corazón, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario de Toledo, Toledo
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Arnau de Vilanova de Valencia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org